CLINICAL TRIAL: NCT03686735
Title: How to Measure Patient Satisfaction
Brief Title: Patient Satisfaction Scales
Status: Completed | Type: Observational
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, David Ring, Associate Dean for Comprehensive Care. Professor of Surgery and Psychiatry, University of Texas at Austin
Other Study IDs: 2018-04-0039
Record Dates: First submitted 2018-08-09; First posted 2018-09-27 (Actual); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: All Orthopedic Disorders; New or Follow-up Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Satisfaction measure 1: 25% of the cohort
  Interventions: Other: 5 anchors and numbers
- Satisfaction measure 2: 25% of the cohort
  Interventions: Other: 5 anchors and no numbers
- Satisfaction measure 3: 25% of the cohort
  Interventions: Other: Visual analog scale with 3 anchors and numbers
- Satisfaction measure 4: 25% of the cohort
  Interventions: Other: Visual analog scale with 3 anchors and no numbers

INTERVENTIONS:
Other: 5 anchors and numbers — How helpful was this visit? 0 This visit was not helpful at all
  1 2-3 There were many ways it could have been better 4 5 Neither useless nor helpful visit 6 7-8 Exceptionally helpful visit 9 10 One of the most helpful doctor visits I have ever had
  Groups: Satisfaction measure 1
Other: 5 anchors and no numbers — How helpful was this visit? This visit was not helpful at all There were many ways it could have been better Neither useless nor helpful visit Exceptionally helpful visit One of the most helpful doctor visits I have ever had
  Groups: Satisfaction measure 2
Other: Visual analog scale with 3 anchors and numbers — How helpful was this visit? 0 neutral/50 100 Least helpful visit Most helpful visit
  Groups: Satisfaction measure 3
Other: Visual analog scale with 3 anchors and no numbers — How helpful was this visit?
  This visit was not Neither useless nor One of the most helpful doctor helpful at all helpful visit visits I have ever had
  Groups: Satisfaction measure 4

SUMMARY:
This study aims to assess differences between 4 types of single satisfaction measures. Secondly, if there is a difference in satisfaction between English speaking and Spanish speaking patients.

ELIGIBILITY:
Inclusion criteria:

* All new or return patients seeing a UE / LE surgeon
* Age 18-89
* Able to provide informed consent
* English speaking
* UT Health Austin Musculoskeletal Institute, Austin Regional Clinic, Seton Institute for Plastic and Reconstructive Surgery, Orthopaedic Specialists of Austin, Texas Orthopedics, and ATX Ortho.

Exclusion criteria:

* Not fluent in English

Ages: 18 Years to 89 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All new and follow-up patients seeing an upper- or lower-extremity surgeon will be invited to enroll at the end of their visit.
Sampling Method: Probability Sample
Enrollment: 256 (Actual)
Dates: Start 2018-06-22 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-02 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction scale 1 | Immediately after the visit. Through study completion, approximately 6 months.
  How helpful was this visit? Scale 1 has 5 anchors and numbers
  Scored from 0-10:
  0 This visit was not helpful at all
  1 2-3 There were many ways it could have been better 4 5 Neither useless nor helpful visit 6 7-8 Exceptionally helpful visit 9 10 One of the most helpful doctor visits I have ever had
  Higher scores indicate more satisfaction
Patient satisfaction scale 2 | Immediately after the visit. Through study completion, approximately 6 months.
  How helpful was this visit? Scale 2 has 5 anchors and no numbers visible for the participant
  Scored from 0-10:
  0 This visit was not helpful at all There were many ways it could have been better Neither useless nor helpful visit Exceptionally helpful visit 10 One of the most helpful doctor visits I have ever had
  Higher scores indicate more satisfaction
Patient satisfaction scale 3 | Immediately after the visit. Through study completion, approximately 6 months.
  How helpful was this visit? Scale 3 is a visual analog scale with 3 anchors and numbers
  Scored from 0-100:
  0 Least helpful visit 50 neutral 100 Most helpful visit
  Higher scores indicate more satisfaction
Patient satisfaction scale 4 | Immediately after the visit. Through study completion, approximately 6 months.
  How helpful was this visit? Scale 4 is a visual analog scale with 3 anchors and no numbers visible for the participant
  Scored from 0-100:
  0 This visit was not helpful at all 50 Neither useless nor helpful visit 100 One of the most helpful doctor visits I have ever had
  Higher scores indicate more satisfaction

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Austin Regional Clinic, Austin, Texas
  - Texas Orthopedics, Austin, Texas
  - HTB Musculoskeletal Institute, Austin, Texas
  - Seton Institute for Plastic and Reconstructive Surgery, Austin, Texas
  - Orthopedic Specialists of Austin, Austin, Texas
  - ATX Ortho, Austin, Texas

IPD SHARING:
Plan to Share IPD: No